CLINICAL TRIAL: NCT05091242
Title: The PREVENT AGITATION Trial II - Children ≤1 Year
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Arash Afshari, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20200708; 2020-005409-26 (EudraCT Number)
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Emergence Delirium
Keywords: Anesthesia; Clonidine; Sevoflurane; Pharmacokinetics; Postoperative Nausea and Vomiting; Postoperative Pain; Infant
MeSH Terms: conditions — Emergence Delirium; Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Clonidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Part A: Open-label pharmacokinetic part (n =16) Part B: Randomized placebo-controlled part (n =320)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clonidine (Experimental): Participants receive Clonidine solution for injection, 3 microg/kg, administered intravenously once over 2 minutes approximately 20 minutes before end of procedure. Injection is administered from a dilated solution of Clonidine 15 microg/mL (ie., 0.2 mL/kg).
  Interventions: Drug: Clonidine
- Placebo (Placebo Comparator): Participants receive Sodium Chloride isotonic (9mg/mL) solution for injection administered intravenously once over 2 minutes approximately 20 minutes before end of procedure. Dosage is administered according to weight: 0.2 mL/kg.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Clonidine — Clonidine injection 3 mcg/kg once
  Other Names: Catapresan; Catapres
  Arms: Clonidine
Drug: Sodium chloride — Sodium chloride 0.9 % injection 0.2 mL/kg once
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Emergence agitation is a clinical condition in which the child experiences a variety of behavioural disturbances including crying, thrashing, and disorientation during early awakening from anaesthesia. Emergence agitation is a common challenge in children with a reported incidence of approximately 25% ranging from 10 to 80 %. Clonidine is often used off-label in paediatric anaesthesia e.g. sedation in the intensive care unit, prevention of withdrawal symptoms after long-term sedation, as premedication before induction of anaesthesia or as treatment/prevention of emergence agitation. The study is designed as a randomised, placebo-controlled clinical trial evaluating efficacy and safety of a single dose of intraoperative clonidine in children 3-12 months, including pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients (male and female), aged 3- ≤ 12 months
* Scheduled general anaesthesia with sevoflurane and opioid. Induction with propofol is optional
* The legally acceptable representative for the study participant provides written informed consent/assent for the trial

Exclusion Criteria:

* ASA >2
* Cardiac, neuro and trauma surgery
* Ex-premature (<37 weeks) • Premedication with clonidine
* Intubated prior to scheduled anaesthesia or is expected to require intubation after the procedure
* Critical illness incl. hemodynamic instability (inotropic drugs needed)
* Bleeding requiring transfusion prior to scheduled anaesthesia
* Planned for a postoperative nurse-controlled analgesia pump including a continuous infusion of opioid
* Malignant disease
* Cardiac disease incl. arrhythmia
* Chronic lung disease that may influence study results or study participation in the opinion of the Investigator or may comprise safety and well-being of the patient
* Mental retardation
* Neurological disease including symptoms similar to emergence agitation
* Has or is suspected of having a family or personal history of malignant hyperthermia
* Has or is suspected of having an allergy to study treatment or its excipients
* Any condition that can in opinion of the Investigator, deteriorate safety and well-being of the patients or interfere with pharmacokinetic data
* Positive Covid-19 test or clinical suspicion of Covid-19 (according to current local guidelines)

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 336 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence agitation during stay in postanaesthetic care unit (PACU) | From admission to PACU to discharge from PACU, up to app. 4 hours. Emergence agitation is considered present ("Yes"), if Watcha score>2 at ANY time point within the given time frame.
  Participants will be assessed on Watcha scale (1=calm, 4=agitated and thrashing around) every 15 minutes from arrival to PACU till discharge therefrom. Emergence agitation is defined dichotomously as Yes/No, Yes being if any Watcha score >2.
Compartmental clearance for pharmacokinetic profiling. | Samples will be collected at baseline and at 5, 15, 30, and 60 minutes post dosage and just prior prior to removal of iv-access ie., at latest 120-240 min post dosage.
  Pharmacokinetic sampling will be performed in 1 mL EDTA tubes and analysed for clonidine plasma concentration in migrog/L
Volume of distribution for pharmacokinetic profiling. | Samples will be collected at baseline and at 5, 15, 30, and 60 minutes post dosage and just prior prior to removal of iv-access ie., at latest 120-240 min post dosage.
  Pharmacokinetic sampling will be performed in 1 mL EDTA tubes and analysed for clonidine plasma concentration in migrog/L
T1/2 for pharmacokinetic profiling. | Samples will be collected at baseline and at 5, 15, 30, and 60 minutes post dosage and just prior prior to removal of iv-access ie., at latest 120-240 min post dosage.
  Pharmacokinetic sampling will be performed in 1 mL EDTA tubes and analysed for clonidine plasma concentration in migrog/L

SECONDARY OUTCOMES:
Proportion of participants with postoperative pain | From admission to PACU to discharge from PACU, up to app. 4 hours.
  Participants will be assessed on Faces Legs Activity Cry Consolability (FLACC) scale every 15 minutes from arrival to PACU till discharge therefrom. Postoperative pain is defined as any FLACC score > 3 during PACU stay.
Proportion of participants with Postoperative Nausea and Vomiting (PONV) | From admission to PACU to discharge from PACU, up to app. 4 hours.
  Participants will be assessed for PONV every 15 minutes during PACU stay. No validated scale for assessment of PONV exists in this age group and PONV will be assessed by dichotomously as "Yes" or "No". While vomiting is obvious, nausea may be considered if participant refuses to eat and other causes are ruled out.
Safety and tolerability of clonidine in infants 3-12 months of age: proportion of participants with adverse events of clinical interest | From administration of intervention through end of anaesthesia and PACU stay (up to app. 4 hours). Supplemental Adverse Event follow-up at 24 hours, 48 hours in case of ongoing adverse events and at 30 days post-intervention.
  Composite outcome combining as assessed by investigator for each participant any clinically relevant hypotension (ie., necessitating intervention), clinically relevant bradycardia (ie., necessitating intervention), clinically relevant apnoea (ie., unexplained cessation of breathing for 20 seconds or longer, or a shorter respiratory pause associated with bradycardia, cyanosis, and/or marked hypotonia).
Mean sedation level in PACU | From admission to PACU to discharge from PACU, up to app. 4 hours.
  Participants will be assessed for alertness on the University of Michigan Sedation Scale (UMSS) every 15 minutes during PACU stay.
Mean amount of additional opioid administered in PACU | From admission to PACU to discharge from PACU, up to app. 4 hours.
  The opioid sparing effect will be evaluated by assessing the amount of additional opioid administered to each participant for postoperative pain during the PACU stay calculated as morphine equivalents.
Mean time to administration of opioid i PACU | From admission to PACU to discharge from PACU, up to app. 4 hours.
  Time in minutes to first administration of opioid will be assessed for each participant during PACU stay.
Mean time to postoperative feeding/oral intake | From admission to PACU to discharge from PACU, up to app. 4 hours.
  Time in minutes from administration of intervention to first time point at which participant is eating during PACU stay, evaluated every 15 minutes.
Mean time to awakening | From admission to PACU to discharge from PACU, up to app. 4 hours.
  Time in minutes from administration of intervention to time point at which participant is awake in PACU, evaluated every 15 minutes. If child is not awake 2 hours after arrival, an awakening attempt will be initiated.
Mean time to discharge readiness | From admission to PACU to discharge from PACU, up to app. 4 hours.
  Time in hours from arrival in PACU to time point at which participant fulfills local PACU discharge criteria as judged by physician, evaluated every 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Afshari, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No